CLINICAL TRIAL: NCT05389787
Title: Impact of Cerebellar TMS on Brain and Cognitive Functions in Schizophrenia: a Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Hengyi Cao, Associate Professor, Northwell Health
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 22-0171
Record Dates: First submitted 2022-05-12; First posted 2022-05-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia; Cerebellar Function; Condition
MeSH Terms: conditions — Schizophrenia; Disease | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TMS (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham (Sham Comparator)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — The TMS will be administrated using the MagVenture Mag Pro R30 device equipped with a B-70 coil. The FDA-approved iTBS sequence will be applied: 10 bursts of three biphasic pulses at 50 Hz, repeated at 5 Hz, for 10 seconds for a total of 600 pulses, and will be repeated for three times. The total stimulation time is ~10 min per session (day). Patients will receive five sessions (days) of rTMS each week, and the total treatment will last for four weeks.

SUMMARY:
This is a single-site, sham-controlled, randomized trial in a total of 40 subjects between ages 18 and 60 years with schizophrenia. This study will investigate the effects of 4-week rTMS treatment on brain and cognitive functions in patients. Subjects will be randomized to one of the following arms:

Arm 1: Standard of Care (SOC) and active rTMS Arm 2: Standard of Care (SOC) and sham rTMS

Each participant will receive rTMS five days per week, for four consecutive weeks. Functional magnetic resonance imaging (fMRI) scans, clinical assessments, and cognitive tests will be performed at baseline, end of the 2nd week, and end of the 4th week.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 to 60 years of age
2. DSM-V diagnosis of schizophrenia spectrum disorders
3. Competent to provide informed consent

Exclusion Criteria:

1. Lifetime DSM-V diagnosis of an Axis-I disorder other than schizophrenia spectrum disorders
2. Lifetime diagnosis of ataxia or other cerebellar disorders
3. Lifetime diagnosis of mental retardation, dementia, Alzheimer's disease, Parkinson's disease, Huntington's disease, or other neurodegenerative disorders
4. Any active general medical condition or CNS disease which can affect cognition or response to treatment
5. Substance dependence or abuse in the past six months
6. Seizure history
7. TMS within three months or ECT within six months
8. Pregnancy as indicated by self-report
9. MRI contraindications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Cerebellar function | end of 2nd week and 4th week
  Changes of cerebellar connectivity after TMS treatment compared with baseline, as measured by functional magnetic resonance imaging (fMRI)

SECONDARY OUTCOMES:
Cognitive function | end of 2nd week and 4th week
  Changes of scores for the Brief Assessment of Cognition in Schizophrenia (BACS) battery after TMS treatment compared with baseline

OTHER OUTCOMES:
Cerebellum-cognition associations | end of 2nd week and 4th week
  Pearson Correlations between changes of cerebellar connectivity (as measured by fMRI) and changes of cognitive scores (as measured by BACS)

CONTACTS AND LOCATIONS:
Locations (1):
- Zucker Hillside Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No